CLINICAL TRIAL: NCT04864197
Title: Assessment of Keratinized Gingiva With and Without PRF Application in Patients With Dental Implant
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Baghdad (Other)
Responsible Party: Principal Investigator, Hussain Falah Mohsen, dentist (MSc student), University of Baghdad
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: U0005B2O
Record Dates: First submitted 2021-04-24; First posted 2021-04-28 (Actual); Last update posted 2021-04-28 (Actual); Status verified 2021-04

CONDITIONS: Thickening; Gingival
MeSH Terms: conditions — Gingival Hyperplasia

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: Third professional person apply PRF membrane.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- prf group (Experimental): prf membrane placement over implant site for gingival thickening
  Interventions: Biological: platelet rich fibrin
- control group (Experimental): no prf placement
  Interventions: Biological: platelet rich fibrin

INTERVENTIONS:
Biological: platelet rich fibrin — prf membrane placement over implant site for gingival thickening
  Other Names: PRF

SUMMARY:
we used prf with dental implant treatment to find out whether prf has an effect on increasing the soft tissue thickness and keratinized tissue width

DETAILED DESCRIPTION:
Clinical oral implant related research is facing many interesting challenges. One of them is to create and maintain stable soft and hard tissues around osseointegrated oral implants.

It was suggested in a classic study that a minimum of 2 mm of keratinized mucosa (KM) around natural teeth is necessary to maintain gingival health. The lack of a sufficient wide zone of KM has been investigated as a potential contributing factor for peri- implant disease and therefore might influence the long- term success of oral implants.

Various studies have found a negative influence of the absence of KM on plaque accumulation. Oral implants with a narrow zone of KM (<2 mm) frequently exhibit significantly higher plaque scores than those with wider zones of KM. Even a subdivision can be made between KM and attached KM (AKM). A statistically significant higher plaque accumulation and gingival inflammation around implants in the groups with KM <2 mm and AKM <1 mm was observed. However, this could not be confirmed in another study.

Interestingly, the presence of an adequate band of KM adjacent to the implant seems to reduce inflammation, hyperplasia and recession of the marginal peri- implant soft tissues. Furthermore, it might facilitate restorative procedures, improve aesthetics and enable the patient to maintain an adequate oral hygiene without irritation or discomfort.

In particular, in the lower jaw, a scarce amount of KM can be regularly encountered. A reduced height of the alveolar process, due to crestal bone resorption, result in loss of KM due to the reduced distance between the bone crest and "genetically defined" position of the mucogingival line. Notably, in the posterior segments of the lower jaw, a narrow KM might be related to muscle pull, high frenulum attachments and a shallow vestibule.

Today, the golden standard to augment KM is a free gingival graft (FGG) harvested from the palate. The main problem with this technique is the morbidity for the patient as it involves a second surgical site. Reported problems following FGG procedure are pain, change in diet, paresthesia, herpetic lesion, mucocele, arteriovenous shunt and excessive bleeding.

To overcome this problem, different authors have proposed alternative techniques and materials to augment keratinized tissue around teeth and oral implants.

Various studies have substantiated the viability of platelet concentrates on enhancement of osseous and associated tissue healing and PRF is one of the recent innovations of various platelet concentrates.

Platelet- rich fibrin (PRF) is a 2nd generation platelet concentrate, which was introduced by Choukroun et al in 2001. It is obtained by a simple and inexpensive procedure that does not require biochemical blood handling. Its 3- dimensional fibrin network promotes neovascularization, accelerates wound closing and fast cicatricle tissue remodeling. Platelet concentrates are considered a source of autologous growth factors that promote cell migration and proliferation. Given that PRF is produced without using any additive, the fibrin polymerization occurs in a physiological way, resulting in a similar fibrin network as the one formed during natural healing.

Studies show a constant release of growth factors such as PDGF (platelet-derived growth factor) or TGF-b (transforming growth factor) for at least 1 week up to 28 days and proved its accelerating effect on the healing process.

ELIGIBILITY:
Inclusion Criteria:

* Patients greater than 18 years old without systemic diseases and having good oral hygiene (with D1-D3 bone density).

Exclusion Criteria:

* general contraindications to implant surgery.
* patients with a history of severe periodontitis.
* bone augmentation required.
* smokers.
* treated or under treatment with intravenous aminobisphosphonates.
* pregnant or lactating.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2019-12-19 (Actual); Primary Completion 2020-07-15 (Actual); Study Completion 2021-07-15 (Estimated)

PRIMARY OUTCOMES:
measuring gingival thickness | 6 months
  transgingival measurement my endodontic reamer and then using digital vernier to determine the thickness

SECONDARY OUTCOMES:
keratinized tissue width | 6 months
  by using periodontal probe

CONTACTS AND LOCATIONS:
Locations (1):
- College of Dentistry / University of Baghdad, Baghdad, Iraq

IPD SHARING:
Plan to Share IPD: No